CLINICAL TRIAL: NCT03272763
Title: A Development Study to Evaluate a Full-Face Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-225
Record Dates: First submitted 2017-08-30; First posted 2017-09-06 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: After a period of baseline, all enrolled participants will be put on the same trial mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- F&P Toffee mask (Experimental): Participants will be placed on this arm for a total of 14 ± 5 days from Visit two. Participants will be using the trial full-face mask during this treatment arm.
  Interventions: Device: F&P Toffee mask

INTERVENTIONS:
Device: F&P Toffee mask — Trial Full-Face mask which comes with three seal sizes and two headgear sizes.

SUMMARY:
This investigation is designed to evaluate the comfort, ease of use and performance of a trial nasal mask for the treatment of Obstructive Sleep Apnea (OSA) in the home environment.

DETAILED DESCRIPTION:
This investigation is a prospective, non-randomized, non-blinded study. Up to 45 OSA participants who currently use a full-face mask will be recruited.

This study will involve a baseline (Visit One) data gathering with the participant's positive airway pressure (PAP) therapy and their usual mask. This will be followed by the participants being fitted with the trial full-face mask for use in-home (Visit Two).

The participant then will come in to return the mask (Visit Three) and give their feedback on their experience using the mask in home in the form of a structured interview during Visit Three. The maximum amount of time the participants will be exposed to the trial mask in-home will be 14 ± 5 days from Visit Two.

The mask and CPAP (if used from the research pool) will be returned to the institution at the conclusion of the trial and participant will return to their usual mask and therapy device for the treatment of their Obstructive Sleep Apnea.

Neither the investigators nor the participants will be blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* AHI ≥ 5 from the diagnostic night
* Aged 22 and over (FDA defined as default)
* Either prescribed APAP, CPAP or Bi-level PAP for OSA
* Existing Full-Face mask user
* Fluent in spoken and written English

Exclusion Criteria:

* Inability to give informed consent
* Participant intolerant to PAP
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or CO2 retention
* Pregnant or think they may be pregnant

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- California Sleep Solutions, Roseville, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers or institutions. Identifiable participant data will not leave the site and all other data will be de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | F&P Toffee Mask
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Trial Mask Comfort
Description: Comfort comparison of trial mask compared to their usual mask. Determined from custom questionnaires - Subjective
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  Much better | 7
  Better | 13
  Same | 3
  Worse | 12
  Much worse | 3

2. Primary Outcome: Trial Mask Performance - Objective
Description: Performance data recorded from the PAP device comparing leak at baseline compared to with trial mask - Objective
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  Increased leak | 9
  Same leak | 3
  Decreased leak | 9
  N/A | 17

3. Primary Outcome: Trial Mask Performance - Subjective
Description: Seal leak in comparison to their usual mask. Determine from questionnaires - Subjective
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  Much better | 9
  Better | 8
  Same | 10
  Worse | 10
  Much worse | 1

4. Primary Outcome: Trial Mask Usability
Description: Whether the patient got the correct orientation and positioning of mask without help. Usability interview - Subjective
Time Frame: During Visit Two - 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  Both orientation and positioning | 17
  Orientation only | 25
  Neither | 1

5. Primary Outcome: Trial Mask Ease-of-Use
Description: Usability of trial mask compared to usual mask. Determined from questionnaires - Subjective
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  Much better | 7
  Better | 14
  Same | 13
  Worse | 3
  Much worse | 1

6. Secondary Outcome: Mask Leak Data
Description: Leak data recorded from PAP device - Objective
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 20
Participants
  Leak increased | 1
  Leak remained the same | 3
  Leak decreased | 10
  No data | 6

7. Secondary Outcome: Seal Size Determination
Description: Did the sizing tool designed for the trial mask correctly predict which size was best suited for the participant.
Time Frame: 1 day-time appointment (1 hour) during Visit Two
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  Yes | 36
  No | 2

8. Secondary Outcome: Efficacy Data
Description: AHI data recorded from PAP device comparing trial mask use to baseline measurements - Objective
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Toffee Mask
Number analyzed (Participants) | 38
Participants
  AHI increased | 18
  AHI remained the same | 3
  AHI decreased | 14
  No data | 3

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for all participants for 1 year from the date informed consent was obtained.
Arm/Group | F&P Toffee Mask
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 2/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F&P Toffee Mask (N=38)
Nasal congestion and sore (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Facial pressure sore on bridge of nose, sinus infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03272763/Prot_SAP_001.pdf